CLINICAL TRIAL: NCT03093129
Title: Phase II Randomised, Double Blind, Placebo Controlled Trial of Neoadjuvant Artesunate in Stage II/III Colorectal Cancer in Vietnamese Patients
Brief Title: Safety and Effectiveness Study of Pre-operative Artesunate in Stage II/III Colorectal Cancer (NeoART-V)
Acronym: NeoART-V
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The 108 Military Central Hospital (Other Government)
Collaborators: Institute of Tropical Medicine, University of Tuebingen (Other)
Responsible Party: Principal Investigator, Le Huu Song, Associate Professor MD,PhD, The 108 Military Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NeoArt-V
Record Dates: First submitted 2017-03-16; First posted 2017-03-28 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Artesunate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- artesunate (Active Comparator): Patients will receive 200 mg artesunate (Arinate®) per oral (PO) once daily (OD) for fourteen days prior to their planned surgery and then be followed up for 5 years following surgery.
  Interventions: Drug: artesunate
- placebo (Placebo Comparator): Patients will receive matching placebo tablets per oral (PO) once daily (OD) for fourteen days prior to their planned surgery and then be followed up for 5 years following surgery.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: artesunate — Artesunate (Trade name : Arinate®)
  Artemisinins are a family of sesquiterpene trioxane anti-malarial agents derived from Sweet wormwood (Artemisia annua L) that have been used in traditional Chinese medicine for centuries to treat fevers. Artesunate, artemether and arteether are derivatives of artemisinin that are converted into their active metabolite dihydroartemisinin (DHA). Artesunate is approved for the treatment of uncomplicated and multidrug-resistant malaria and is on the WHO list of Essential Medicines (WHO., 2015).
  Other Names: Arinate®
  Arms: artesunate
Other: placebo — The matching placebo tablets contain lactose monohydrate, microcrystalline cellulose, croscarmellose sodium, colloidal anhydrous silica and a magnesium stearate blend.
  Arms: placebo

SUMMARY:
This is a Phase II randomized, double-blind, placebo-controlled trial of neoadjuvant artesunate given orally as a dose of 200 mg once a day for 14 days to patients with histologically confirmed Stage II/III colorectal cancer (CRC) awaiting surgical treatment with curative intent.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer worldwide and represents a significant health care burden with an incidence of one million new cases per year. In Vietnam, Colorectal cancer is the third most common cause of cancer deaths in men and fourth in women. Artesunate is a safe and effective antimalarial with evidence of anticancer properties across a range of cancer cell lines. Results from a pilot feasibility study in colorectal cancer patients in the UK showed that artesunate was safe and well tolerated. These findings provided the basis for a Phase II clinical trial investigating the effects of neoadjuvant artesunate on progression free survival and overall survival in Stage II/III Colorectal Cancer in Vietnamese Patients.

Artesunate given orally as a dose of 200 mg once a day for 14 days to patients with histologically confirmed Stage II/III colorectal cancer (CRC) awaiting surgical treatment with curative intent.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Histologically proven single primary site colorectal adenocarcinoma
* Stage II/III colorectal cancer planned for surgical resection and no clinical indication for neoadjuvant preoperative chemotherapy/chemoradiation therapy
* WHO performance status 0,1 or 2
* Adequate full blood count: White Cell Count (WCC) >3.0 x 109 /l; Platelets >100 x 109/l; Haemoglobin (Hb) >8g/dL
* Adequate renal function : Glomerular Filtration Rate >30ml/min by Cockcroft-Gault formula
* Adequate hepatobiliary function : Bilirubin < 3 x Upper limit normal
* Female participants of child bearing potential must have a negative pregnancy test < 72 hours prior to initiating study intervention and agree to avoid pregnancy using contraceptive precautions for up to 6 weeks after the last dose of study treatment intervention
* Male participants with a partner of childbearing potential must agree to use contraceptive precautions during and for up to 6 weeks after the last dose of the study treatment intervention
* Patient able and willing to provide written, informed consent for the study

Exclusion Criteria:

* Contraindication to the use of artesunate due to hypersensitivity
* Pregnancy or lactation
* History of immunosuppression
* History of hearing or balance problems
* Weight < 42 kg or > 110 kg
* Other planned intervention, apart from Vietnamese standard of care
* Any other malignant disease diagnosis within the preceding 2 years with the exception of non-melanomatous skin cancer and carcinoma in situ
* Lactose intolerance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
recurrence free survival 2 years after surgery | 2 years
  The primary outcome measure for the comparison of the artesunate versus placebo group is recurrence free survival 2 years after surgery

SECONDARY OUTCOMES:
Recurrence free survival at 5 years | 5 years
  Recurrence free survival
Overall survival at 2 and 5 years | 2-5 years
  Overall survival
Colon cancer specific death at 2 and 5 years | 2-5 years
  Colon cancer specific death
Artesunate drug related toxicity | 5 years
  drug related toxicity
Pathological assessment of tumour regression (involvement of lymph nodes ; serosa ; resection margin) | 5years
  Pathological assessment
Surgical morbidity/mortality | 5years
  Surgical morbidity/mortality
Predictive value of tumour biomarkers in terms of predicting response to artesunate therapy | 5 years
  tumour biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Mai Hong Bang, MD,PhD, Study Director — 108 Military Central Hospital
Locations (1):
- 108 Military Central Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Krishna S, Ganapathi S, Ster IC, Saeed ME, Cowan M, Finlayson C, Kovacsevics H, Jansen H, Kremsner PG, Efferth T, Kumar D. A Randomised, Double Blind, Placebo-Controlled Pilot Study of Oral Artesunate Therapy for Colorectal Cancer. EBioMedicine. 2014 Nov 15;2(1):82-90. doi: 10.1016/j.ebiom.2014.11.010. eCollection 2015 Jan. PMID 26137537